CLINICAL TRIAL: NCT00759811
Title: METhotrexate Therapy Effects in the Physical Capacity of Patients With ISchemic Heart Failure: Randomized Double-blind, Placebo-controlled Trial (METIS Trial)
Brief Title: METhotrexate Therapy Effects in the Physical Capacity of Patients With ISchemic Heart Failure (METIS Trial)
Acronym: METIS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Daniel Medeiros Moreira, MSc., Instituto de Cardiologia do Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: UP4062
Record Dates: First submitted 2008-09-24; First posted 2008-09-25 (Estimated); Results first posted 2013-05-08 (Estimated); Last update posted 2013-05-08 (Estimated); Status verified 2013-03

CONDITIONS: Heart Failure; Myocardial Ischemia
Keywords: Heart Failure; Myocardial Ischemia; Methotrexate; Inflammation; Anti-Inflammatory Agents; Inflammation Mediators
MeSH Terms: conditions — Heart Failure; Myocardial Ischemia; Inflammation | interventions — Methotrexate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Methotrexate (Experimental): Patients receiving conventional treatment to heart failure who will receive methotrexate 7.5mg oral plus folic acid 5mg oral once a week for 12 weeks.
  Interventions: Drug: Methotrexate
- Placebo (Placebo Comparator): Patients receiving conventional treatment to heart failure who will receive placebo oral plus folic acid 5mg oral once a week for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methotrexate — Patients receiving conventional treatment to heart failure who will receive methotrexate 7.5mg oral plus folic acid 5mg oral once a week for 12 weeks.
  All patients will have evaluated at the baseline and after 12 weeks: physical capacity by the 6-minutes walk test, quality of life by the Brazilian edition SF-36 and inflammatory marker by C-reactive protein. They also will be tested for ALT, AST, blood cell count, creatinine, and prothrombin time at baseline, after 6 weeks and after 12 weeks.
  Other Names: Rheumatrex; Trexall
  Arms: Methotrexate
Drug: Placebo — Patients receiving conventional treatment to heart failure who will receive placebo oral plus folic acid 5mg oral once a week for 12 weeks.
  All patients will have evaluated at the baseline and after 12 weeks: physical capacity by the 6-minutes walk test, quality of life by the Brazilian edition SF-36 and inflammatory marker by C-reactive protein. They also will be tested for ALT, AST, blood cell count, creatinine, and prothrombin time at baseline, after 6 weeks and after 12 weeks.
  Other Names: Control
  Arms: Placebo

SUMMARY:
The aim of the study is to evaluate the efficacy of methotrexate to improve physical capacity in patients with symptomatic ischemic heart failure.

DETAILED DESCRIPTION:
Recent studies have showed the importance of proinflammatory mediators in the heart failure. However, there is a lack of benefit of therapies that tried to neutralize these mediators.

Methotrexate has adenosine-mediated anti-inflammatory effects in rheumatoid arthritis and psoriasis. Methotrexate limits infarct size via this adenosine-dependent mechanisms in heart of dogs (J Cardiovasc Pharmacol. 2004 Apr;43(4):574-9). A recent trial showed that this drug reduced proinflammatory mediators in patients with heart failure (Am Heart J. 2006 Jan;151(1):62-8).

These data suggest that methotrexate may improve physical capacity in patients ischemic heart failure reducing inflammation, but a randomized clinical trial is necessary to prove it.

ELIGIBILITY:
Inclusion Criteria:

* Heart failure functional class measured using the New York Heart Association classification class II, III or IV
* Left ventricular fraction <0.45 at the ventriculography
* Angiographic coronary lesions higher than 50% or coronary lesion revascularized (coronary artery bypass or percutaneous transluminal coronary angioplasty)

Exclusion Criteria:

* Myocardial infarction in the past four months
* Coronary artery bypass or percutaneous transluminal coronary angioplasty in the past four months
* Left ventricular disfunction diagnosed during a acute coronary syndrome
* Those who require revascularization in the following 12 weeks
* Hepatic disease (ALT and AST higher than the upper limit of the reference value)
* Renal failure (plasma creatinine higher than 2.0mg/dl)
* Alcoholism (20 doses per week or more)
* Illegal drug use
* Rheumatoid arthritis or other inflammatory diseases
* Infectious disease
* Neoplasm
* Anemia (hematocrit lower than 30%)
* Currently on any anti-inflammatory drugs
* Difficulty in walking
* Unable to understand/complete the 36-item Short Form health survey (SF-36)
* Those who do not give informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2007-12; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Carlos AM Gottschall, MD MSc PhD, Study Director — Instituto de Cardiologia do Rio Grande do Sul; Daniel M Moreira, MD, Principal Investigator — Instituto de Cardiologia do Rio Grande do Sul; Jefferson L Vieira, MD, Study Director — Instituto de Cardiologia do Rio Grande do Sul
Locations (1):
- Instituto de Cardiologia do Rio Grande do Sul / Fundação Universitária de Cardiologia, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Result] Moreira DM, Vieira JL, Gottschall CA. The effects of METhotrexate therapy on the physical capacity of patients with ISchemic heart failure: a randomized double-blind, placebo-controlled trial (METIS trial). J Card Fail. 2009 Dec;15(10):828-34. doi: 10.1016/j.cardfail.2009.06.439. Epub 2009 Aug 5. PMID 19944358

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Methotrexate | Placebo
Started | 25 | 25
Completed | 23 | 24
Not Completed | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Methotrexate | Placebo | Total
Number analyzed (Participants) | 25 | 25 | 50
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 16 | 18 | 34
  >=65 years | 9 | 7 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 60.8 (10.3) | 58.2 (8.0) | 59.5 (9.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 4 | 11
  Male | 18 | 21 | 39
Region of Enrollment [Number; unit: participants]
  Brazil | 25 | 25 | 50

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Capacity Measured Using the 6-minute Walk Test Distance
Description: The primary outcome of the study was the difference in 6MWT distance before and after the treatment (change in meters evaluated by t test).
Time Frame: Baseline and 12 weeks
Measure: Mean (Standard Deviation); unit: meters
Arm/Group | Methotrexate | Placebo
Number analyzed (Participants) | 25 | 25
meters | 24.5 (39.5) | 21.3 (43.7)

2. Secondary Outcome: Improve in Heart Failure Functional Class Measured Using New York Heart Association
Time Frame: 12 weeks
Reporting Status: Not Posted

3. Secondary Outcome: Improve in Quality of Life Measured Using the Brazilian Edition SF-36
Time Frame: 12 weeks
Reporting Status: Not Posted

4. Secondary Outcome: Reduction of Inflammatory Marker Measured Using C-reactive Protein Blood Levels
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Incidence of All Cause Mortality, Hospitalization for Worsening Heart Failure, Myocardial Infarct, Stroke or Myocardial Revascularization Need
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Incidence of Adverse Effects of the Treatment
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Methotrexate | Placebo
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/24
Other Adverse Events (participants affected / at risk) | 7/23 | 9/24
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Methotrexate (N=23) | Placebo (N=24)
nausea (Gastrointestinal disorders) | 2 | 2
lipothymia (Nervous system disorders) | 1 | 2
sustained ventricular tachycardia (Cardiac disorders) | 1 | 0
dizziness (Nervous system disorders) | 3 | 5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes